CLINICAL TRIAL: NCT02055690
Title: A Phase Ib and Randomised Phase II Trial of Pazopanib With or Without Fosbretabulin in Advanced Recurrent Ovarian Cancer
Brief Title: PAZOFOS: Phase Ib and Phase II Trial of Pazopanib +/- Fosbretabulin in Advanced Recurrent Ovarian Cancer
Acronym: PAZOFOS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Safety
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Novartis (Industry); Mateon Therapeutics (Industry); East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13_DOG01_119; 2013-005471-40 (EudraCT Number)
Record Dates: First submitted 2014-02-02; First posted 2014-02-05 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Ovarian Neoplasms; Neoplasms, Ovarian; Ovarian Cancer
Keywords: Advanced Recurrent Ovarian Cancer; Pazopanib; Votrient; Fosbretabulin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pazopanib; fosbretabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase Ib/II: Fosbretabulin & Pazopanib (Experimental): Phase Ib:
  Fosbretabulin and Pazopanib in combination. Fosbreatabulin dose will be in the range of 45mg/m2- 60 mg/m2 delivered by infusion every week for 3 weeks of a 4 week cycle until disease progression. Pazopanib will be either 600 mg or 800mg taken orally each day of 28 day cycle until disease progression.
  The phase II dose of both drugs will be determined by the Phase Ib component which is a dose finding exercise.
  Phase II:
  Fosbretabulin and Pazopanib in combination. Fosbretabulin 54mg/m2 delivered by infusion every week for 3 weeks of a 4 week for 28 day cycle until disease progression. Pazopanib 600mg taken orally each day for 28 day cycle until disease progression
  Interventions: Drug: Pazopanib; Drug: Fosbretabulin
- Phase II: Pazopanib (Active Comparator): Pazopanib 800mg taken orally each day of 28 day cycle until disease progression
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Tyrosine Kinase Inhibitor
  Other Names: Votrient; EU/1/10/628/001; EU/1/10/628/002
Drug: Fosbretabulin — Vascular Disrupting Agent
  Other Names: Fosbretabulin tromethamine
  Arms: Phase Ib/II: Fosbretabulin & Pazopanib

SUMMARY:
The first part of this study is to find the recommended dosages of a combination of two drugs: pazopanib and fosbretabulin, which will be given to female patients with relapsed ovarian cancer.

The second part of the study involves comparing the recommended dose of pazopanib and fosbretabulin in combination against pazopanib alone in female patients with relapsed ovarian cancer to determine whether the combination is more beneficial that pazopanib on it's own.

DETAILED DESCRIPTION:
Ovarian cancer is the fourth biggest contributor to female cancer mortality, accounting for 4% of all malignancies diagnosed in women. In the United Kingdom (UK), there are seven thousand new cases of ovarian cancer annually and four thousand two hundred deaths from the disease. The standard treatment approach currently consists of surgical debulking and chemotherapy, usually based around a combination of carboplatin and paclitaxel. Most ovarian cancers are initially chemo-responsive however the majority of patients whose disease initially responds subsequently develop recurrent disease.

Once patients recur, treatment options become less numerous and less effective. Progression free survival rates for platinum-sensitive disease are only about 13 months and the outlook for patients with platinum-resistant disease is much worse.

This study is exploring a new combination of drugs fosbretabulin, a vascular disrupting agent and pazopanib, a tyrosine kinase inhibitor. There is scientific rational for combining these two types of drugs as they should be able to work in combination through contrasting mechanisms of action.

The first part of the study is a dose finding exercise with cohorts of patients being given drugs with in combination until the recommended dose of both drugs is found. Patients in each cohort will be monitored closely for safety and drug toxicity.

The second part of the study has a randomised component where patients will receive the combination of drugs or pazopanib alone with the aim to determine whether there is an advantage in progression free survival for patients that receive pazopanib and fosbretabulin. This will be monitored by RECIST.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, progressive, recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma, which has recurred following at least one platinum-containing regimen.
* Progressive disease according to RECIST 1.1 or GCIG criteria within 3-12 months of completing platinum containing therapy, although this need not be the immediately preceding regimen.
* World Health Organisation (WHO) performance status of 0 or 1 (Appendix 1).
* Measurable disease (RECIST 1.1 (Appendix 2) or Progressive Disease (PD) according to CA125 GCIG criteria with non-measurable disease on CT scan.
* Life expectancy of at least 12 weeks.
* Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient receives the first dose of Investigational Medicinal Product (IMP):

  * Haemoglobin (Hb) ≥ 90 g/L
  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Serum potassium within normal range
  * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≤ 2.5 x ULN unless raised due to hepatic metastatic disease in which case up to 5 x ULN is permissible
  * Either: Calculated creatinine clearance ≥ 40 mL/min (uncorrected value) Or: Isotope clearance measurement ≥ 40 mL/min (corrected)
  * Activated partial thromboplastin time (aPTT) ≤ 1.2 x ULN
  * Prothrombin Time (PT) or International normalised ratio (INR) ≤ 1.3 x ULN
  * Urine protein dipstick of less than or equal to 2+, or if 2+ or greater the patient must have a 24 hour urinary protein value of less than 2 g.
  * Clinically euthyroid.
  * Aged 18 years or over at the time of consent.
  * Written (signed and dated) informed consent and capable of co-operating with treatment and follow-up.
  * Patients can have received bevacizumab prior to trial entry providing that the last dose was administered at least 6 months before the first dose of IMP.

Exclusion Criteria:

* Radiotherapy, surgery or tumour embolisation within 28 days before the first dose of IMP
* Endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C and six weeks for investigational medicinal products) before the first dose of IMP.
* Ongoing grade ≥ 2 toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Chief and Principal Investigators should not exclude the patient; and grade 1 or 2 neurotoxicity considered to be due to paclitaxel.
* Female patients who are able to become pregnant (or are already pregnant or lactating). Those who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
* Major thoracic or abdominal surgery from which the patient has not yet recovered.
* At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
* Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* History of any of the following cardiovascular conditions within the last six months:

  * Coronary revascularisation (percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG))
  * Acute coronary syndrome (myocardial infarction (MI), unstable angina)
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) (Appendix 4)
* Patients who have sustained hypertension, defined as a systolic blood pressure (SBP) of > 140 mm Hg or diastolic blood pressure (DBP) of > 90 mm Hg, on three occasions.
* ECG with evidence of clinically significant abnormalities.
* Patients with a QTc> 480ms or taking any drug known to prolong the QTc interval that cannot be stopped for the duration of the trial (Appendix 4).
* Patients with pathologic bradycardia (<60 b/m in non-athletes), heart block (excluding first-degree block, being PR interval prolongation only).
* History of cerebrovascular accident (including transient ischaemic attack (TIA)), pulmonary embolism or untreated deep vein thrombosis (DVT) within the past six months. Patients with recent DVT or pulmonary embolism who have been treated with therapeutic anti-coagulant agents for at least six weeks will be eligible, provided their INR (if taking oral anti-coagulants) has been stable for this period of time.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic and have had no requirement for steroids or anti-convulsant medication for six months prior to the first dose of IMP.
* Clinically significant abnormalities that may increase the risk of gastrointestinal bleeding or perforation, including but not limited to:

  * Bleeding: Active peptic ulcer disease, known intraluminal metastatic lesions with risk of bleeding, Inflammatory bowel disease (Crohn's disease, ulcerative colitis);
  * Perforation: History of abdominal fistula or large pelvic mass; gastrointestinal perforation or intra-abdominal abscess within four weeks prior to first dose of IMP; previous bowel surgery which is judged by the investigator to increase significantly the risk of gastrointestinal complications from trial treatment
* Evidence of active bleeding or bleeding diathesis.
* Transfusion within one week prior to first dose of IMP.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
* Clinically significant haemoptysis, within eight weeks before the first dose of IMP.
* Previous treatment with pazopanib.
* Any participant that is participating in (or plans to participate in) another interventional clinical trial, whilst taking part in this Phase Ib/II study of fosbretabulin and pazopanib. Participation in an observational trial would be acceptable.
* Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin and no evidence of recurrence of other malignancy for at least 2 years.
* Hypersensitivity to Pazopanib or any of it's excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Dose Limiting Toxicities of Dose of Pazopanib and Fosbretabulin | 4 weeks after starting treatment (1 cycle)
  To determine the dose of Pazopanib and Fosbretabulin in combination by recording Dose Limiting Toxicities (DLTs) at each cohort level as categorised by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Assessment of toxicity will take place over the 4-week period that constitutes one cycle
Phase II: Progressive disease | Progressive disease (average of 4 months from start of treatment) measured by RECIST
  To determine whether fosbretabulin and pazopanib in combination improves progression free survival compared to pazopanib alone measured by RECIST
  Computed Tomography (CT) scans are taken every 8 weeks for the first 6 cycles and evaluated by the Response Evaluation Criteria In Solid Tumours (RECIST) criteria.
  After 6 cycles of fosbretabulin and pazopanib patients will receive pazopanib alone and CT scans will be undertaken every 3 months (12 weeks).

SECONDARY OUTCOMES:
Phase I: Biomarker changes on a cohort-by cohort basis | Samples taken within the 4 weeks prior to the first dose of drug and during first cycle (weeks 2 and 3) and then at progressive disease (average of 4 months from start of treatment)
  Circulating markers of angiogenesis: VEGFA (Vascular Endothelial Growth Factor), VEGFR2, Ang1 (Angiopoietin), Ang2 and Tie (Tyrosine kinase with immunoglobulin-like and EGF-like domains) 2 will be measured from samples taken pre-treatment and during cycle 1 of treatment
Phase Ib and Phase II: Safety and Toxicity profile of Pazopanib and Fosbretabulin in combination | Adverse Events recorded within the 4 weeks prior to the first dose of drug is administered and during the first 3 weeks of a 4 week cycle of treatment for 6 cycles, then every month until progressive disease (average of 4 months from start of treatment)
  The Phase Ib component is estimated to last approximately 9 months with the total duration of the trial expected to last 45 months. All adverse events will be recorded and categorised by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
  Patients will receive up to six cycles of fosbretabulin and pazopanib after which treatment will be continued with pazopanib alone until progressive disease. It is estimated each patient will be on the trial for approximately 4 months.
Phase II: Biomarker signature for Progression Free Survival | Samples taken within the 4 weeks prior to first dose of drug
  To investigate whether the pre-treatment biomarker signature can predict which patients have a response and a longer progression free survival
  Circulating markers of angiogenesis: VEGFA, VEGFR2, Ang1, Ang2 and Tie 2 will be measured by ELISA and compared to progression free survival data
Phase II: Response rates by RECIST and GCIG CA-125 criteria | Progressive disease (average of 4 months from start of treatment) measured by RECIST and CA125 biomarkers
  The response rate in the pazopanib and combination arms according to RECIST and Gynaecologic Cancer Intergroup (GCIG) Cancer Antigen 125 (CA-125) criteria
  CT scans every every 8 weeks for the first 6 cycles then every 3 months until progressive disease (average of 4 months from start of treatment). CA125 taken twice per cycle for first 6 and then every month until progressive disease
Phase II: Biomarker response in combination arm | Samples taken within the 4 weeks prior to the first dose of drug, Cycle 1 (weeks 2 and 3) and at progression (average of 4 months from start of treatment)
  To investigate whether biomarkers can demonstrate additivity of the combination in comparison with single agent pazopanib
  Circulating markers of angiogenesis: VEGFA, VEGFR2, Ang1, Ang2 and Tie 2 will be measured from samples taken pre-treatment and during cycle 1 of treatment and at progression.
  Circulating endothelial progenitor cells (CEPCs) from these samples will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, Study Chair — The Christie National Health Service (NHS) Foundation Trust; Gordon Rustin, Study Chair — East and North Herts NHS Trust
Locations (10):
- United Kingdom (10):
  - Royal United Hospital Bath NHS Trust, Bath
  - City Hospital, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University Collage London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Metropolitan Borough of Wirral
  - Mount Vernon Cancer Centre (East and North Herts NHS Trust), Middlesex
  - Freeman Hospital (Newcastle-upon-Tyne Hospitals NHS Foundation Trust), Newcastle upon Tyne
  - Oxford Radcliffe Hospitals NHS Trust, Oxford

REFERENCES:
- [Derived] Morgan RD, Banerjee S, Hall M, Clamp AR, Zhou C, Hasan J, Orbegoso C, Taylor S, Tugwood J, Lyon AR, Dive C, Rustin GJS, Jayson GC. Pazopanib and Fosbretabulin in recurrent ovarian cancer (PAZOFOS): A multi-centre, phase 1b and open-label, randomised phase 2 trial. Gynecol Oncol. 2020 Mar;156(3):545-551. doi: 10.1016/j.ygyno.2020.01.005. Epub 2020 Jan 10. PMID 31932108
- See also: Christie NHS website — http://www.christie.nhs.uk/